CLINICAL TRIAL: NCT01840566
Title: A Phase I Trial of High Dose Therapy and Autologous Stem Cell Transplantation Followed by Infusion of Chimeric Antigen Receptor (CAR) Modified T-Cells Directed Against CD19+ B-Cells for Relapsed and Refractory Aggressive B Cell Non-Hodgkin Lymphoma
Brief Title: High Dose Therapy and Autologous Stem Cell Transplantation Followed by Infusion of Chimeric Antigen Receptor (CAR) Modified T-Cells Directed Against CD19+ B-Cells for Relapsed and Refractory Aggressive B Cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-117
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Relapsed; Refractory; Autologous Stem Cell Transplantation; HIGH DOSE CHEMOTHERAPY; 19-28z T cells/kg; 12-117
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — Carmustine; Etoposide; Cytarabine; Melphalan; pegfilgrastim

ARMS (1):
- HIGH DOSE CHEMOTHERAPY AND ASCT (Experimental): This is a phase 1 dose escalation study designed to determine the maximum tolerated dose (MTD) of CAR modified T cells in patients with relapsed and refractory aggressive B-NHL. Three dose levels (5 x 106 19-28z T cells/kg, 1 x 107 19-28z T cells/kg, and 2 x 107 19-28z T cells/kg) are considered for the MTD.
  Interventions: Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Biological: Pegfilgrastim; Biological: 19-28z T CELLS; Procedure: Autologous Stem Cell Transplantation

INTERVENTIONS:
Drug: Carmustine
Drug: Etoposide
Drug: Cytarabine
Drug: Melphalan
Biological: Pegfilgrastim
Biological: 19-28z T CELLS
Procedure: Autologous Stem Cell Transplantation

SUMMARY:
The purpose of this study is to test the safety of delivering the patients' own immune cells, called T cells, after the high-dose chemotherapy (HDT) and autologous stem cell transplantation (ASCT).

ELIGIBILITY:
Transplant eligible patients will be eligible if criteria met per below.

Inclusion Criteria:

* Patients ≥ 18 years of age with aggressive B-cell non-Hodgkin lymphoma subtypes including, relapsed or refractory diffused large B-cell lymphoma (DLBCL), and transformed follicular lymphoma meeting at least one of the following criteria:

  * Bone marrow involvement at the time of relapse or refractory disease and not appropriate for allogeneic transplantation.
  * PET positive disease outside of one radiation port unless single-port disease treated with prior radiotherapy within the port, following > or = to 2 cycles of salvage chemotherapy, still achieving chemosensitive status 1999 IWG criteria (section 12.2 and 12.383).
* Creatinine ≤ 1.5 mg/100 ml (or measured 24 hour creatinine clearance of ≥ 50 cc/min)
* Bilirubin <2.0 mg/100 ml, AST and ALT <3x the upper-limit of normal, PT and PTT < 2x normal outside the setting of stable chronic anticoagulation therapy,
* Adequate cardiac function (LVEF>40%) as assessed by ECHO or MUGA scan performed within 1 month of treatment.
* Adequate pulmonary function as assessed by DLCO of > or = to 45% adjusted for hemoglobin.
* Life expectancy of > 3 months.

Exclusion Criteria:

* Karnofsky performance status ≤ 70 (see appendix VI).
* Patients with other aggressive B-cell malignancies including, but not limited to: Burkitt lymphoma, transformed CLL/SLL and transformed marginal zone lymphoma that are not included in 6.1 inclusion criteria.
* Patients previously treated with autologous or allogeneic bone marrow or stem cell transplantation are ineligible.
* Other past or current malignancy unless in the opinion of the investigator it does not contraindicate participation in the study.
* Uncontrolled bacterial, viral or fungal infection.
* Patients with HIV, active hepatitis B or hepatitis C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-04; Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 2 years
  will be assessed utilizing a standard 3+3 cell dose escalation to determine the maximum tolerated dose of CD19+ CAR T cells
safety | 2 years
  Toxicity will be graded on a scale of 1 to 5 as described by the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 4.0

SECONDARY OUTCOMES:
2 year progression-free (PFS) | 2 years
overall survival (os) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Craig Sauter, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activites), Rockville Centre, New York

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Sauter CS, Senechal B, Riviere I, Ni A, Bernal Y, Wang X, Purdon T, Hall M, Singh AN, Szenes VZ, Yoo S, Dogan A, Wang Y, Moskowitz CH, Giralt S, Matasar MJ, Perales MA, Curran KJ, Park J, Sadelain M, Brentjens RJ. CD19 CAR T cells following autologous transplantation in poor-risk relapsed and refractory B-cell non-Hodgkin lymphoma. Blood. 2019 Aug 15;134(7):626-635. doi: 10.1182/blood.2018883421. Epub 2019 Jul 1. PMID 31262783
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/